CLINICAL TRIAL: NCT06953258
Title: Effects of Home-Based Eccentric Training at Long Muscle Length on Functional Capacity and Neuromechanical Function in Healthy Older Adults
Brief Title: Effects of Eccentric Training at Long Muscle Length on Functional Capacities of Elderly Adults
Acronym: EMULE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Robin Souron (Other)
Collaborators: Pole Hospitalo-Universitaire de Gérontologie Clinique, CHU de Nantes (Unknown); Agence nationale de la recherche (ANR)see www.agence-nationale-recherche.fr (Unknown)
Responsible Party: Sponsor-Investigator, Robin Souron, Associate professor, Institut Pasteur de Lille
Organization: Institut Pasteur de Lille (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMULE 24.03657.000456
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Eccentric Exercise; Home-based Training; Elderly Adults
Keywords: aging; eccentric training; supervision; functional capacities; neuromechanical properties
MeSH Terms: interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: We will compare two training groups that differ in the way the exercises are performed: one group will perform the eccentric phase of the movement at long muscle length, while the other will complete the same exercises in their conventional form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long muscle length eccentric training program (Experimental): Participants assigned to this arm will complete a home-based training program consisting of 24 sessions, including 20 sessions performed independently at home and 4 sessions conducted in small groups at the laboratory. The laboratory-based sessions will be scheduled in coordination with each participant to ensure regular spacing-approximately one supervised session every five home-based sessions-while accommodating individual availability. Group sizes will be maintained between 2 and 5 participants per session to foster motivation and promote adherence.
  The training program will include conventional resistance exercises, with progressive increases in intensity and volume tailored to each participant's capabilities. In this intervention group, four specific exercises targeting the knee extensors and plantar flexors will be performed at long muscle lengths, distinguishing it from Group #2, where these exercises will be performed in a conventional manner (i.e., at neutral or shorter mus
  Interventions: Other: Home-based eccentric training at long muscle length
- Conventional training program (Active Comparator): Participants in this arm will follow a home-based resistance training program consisting of 24 sessions, including 20 sessions performed independently at home and 4 sessions conducted in small groups at the laboratory, as previously described. The training will involve conventional resistance exercises, with progressive adjustments in intensity and volume based on each participant's physical capacity and progression.
  Note: the total training volume (i.e., number of repetitions × number of sets, in arbitrary units) will be matched between groups, ensuring that any differences in outcomes can be attributed to the specific training modality rather than differences in workload.
  Interventions: Other: Conventional home-based training

INTERVENTIONS:
Other: Home-based eccentric training at long muscle length — The training program will include conventional resistance exercises, with progressive increases in intensity and volume tailored to each participant's capabilities. In this condition, specific to the Arm #1, four specific exercises targeting the knee extensors and plantar flexors will be performed at long muscle lengths.
  Other Names: Physical training
  Arms: Long muscle length eccentric training program
Other: Conventional home-based training — The training program will include conventional resistance exercises, with progressive increases in intensity and volume tailored to each participant's capabilities. In this condition, specific to the Arm#2, four specific exercises targeting the knee extensors and plantar flexors will be performed in a conventional manner (i.e., at neutral or shorter muscle lengths).
  Other Names: Physical training
  Arms: Conventional training program

SUMMARY:
As aging leads to a decline in muscle function and overall physical performance, interventions targeting muscle strength and neuromechanical properties are critical for maintaining functional independence in older adults. Long-length eccentric training has shown promise in enhancing muscle performance, but its effects in older adults, particularly in a home-based setting, remain underexplored.

The aim of this trial is to assess whether a targeted home-based training intervention incorporating long-length eccentric contractions can enhance functional capacity and neuromechanical properties in healthy older adults. Participants will be semi-randomly allocated to one of two groups: an experimental group incorporating long-length eccentric contractions (Group 1) or a conventional resistance training group (Group 2), with group assignment stratified to ensure an equal number of men and women in each group. Each participant will complete three laboratory-based experimental sessions (i.e., two Pre-training sessions and one Post-training session) , during which five key evaluations will be conducted: (i) the 5-Time Sit to Stand test, serving as the primary outcome measure; (ii) the Timed Up and Go test; (iii) assessments of isometric and dynamic muscle strength in the knee extensors and plantar flexors; (iv) measurements of the cross-sectional areas of the vastus lateralis, rectus femoris, gastrocnemius medialis, and soleus muscles; and (v) evaluation of tendon stiffness.

Following the pre-evaluation, each participant will engage in a 24-session, semi-supervised, home-based training protocol over a period of 8 to 11 weeks. The training program will include eight exercises, with four targeting the upper limbs and four focused on the lower limbs. Group 1 will perform the lower limb exercises at long muscle lengths, while Group 2 will perform the same exercises in a conventional manner (i.e., at neutral or shorter muscle lengths). The total training volume (calculated as repetitions × sets, in arbitrary units) will be matched across both groups, ensuring that any observed differences in outcomes are attributable to the specific training modality rather than differences in workload.

DETAILED DESCRIPTION:
Home-based resistance training has emerged as a practical alternative for individuals who lack access to traditional, facility-based exercise programs. This is particularly relevant for older adults, who often face multiple barriers to participating in supervised center-based training-the current gold standard-including reduced mobility, transportation difficulties, and financial constraints. As a result, home-based programs can offer a more accessible option to support engagement in resistance training. Evidence suggests that home-based resistance training can lead to improvements in strength and functional capacity among healthy older individuals; however, these gains tend to be modest. One key limitation is that exercise intensity in home settings may not progress adequately over time, often due to the absence of supervision or limited motivation to increase effort.

Besides training localization and level of supervision, the modality of contraction appears to be of importance. Previous evidences in young but also elderly adults suggest that eccentric training should be performed at long muscle length to obtain the greatest improvements in neuromuscular and physical functions. At the muscle level, the force-length relationship indicates that muscle tension is greater at long vs short muscle length. This is an obvious but important point since mechanical tension during training exercises is a key parameter for muscle plasticity and strength gains. It has been reported positive effects of a short-term (i.e. 3-week) eccentric training performed in a lengthened position on architectural and functional characteristics of the hamstrings in young adults. However, they found no difference between long and short muscle lengths, likely because of the short training duration. It has also been reported significant neuromuscular (e.g. fascicle length, pennation angle, voluntary activation level) and functional (e.g. muscle force) improvements after a 6-week eccentric training at long muscle length in the hamstrings of young adults. Resistance training interventions focusing on eccentric contractions seem particularly interesting for older individuals, as they are less metabolically demanding than concentric contractions for comparable workloads.

Although home-based resistance training programs emphasizing eccentric contractions have been shown to be more effective than those focusing on concentric contractions for improving lower limb strength, mobility, and postural stability in healthy older adults, the integration of eccentric exercises performed at long muscle lengths within home-based protocols has yet to be explored. This represents a significant challenge, as both contraction intensity and muscle length are difficult to monitor and control in real-world, home-based settings compared to tightly controlled laboratory environments.

The aim of this trial is to assess whether a home-based resistance training program incorporating long-length eccentric contractions of the lower limbs can lead to greater improvements in functional capacities and neuromechanical properties in healthy older adults compared to a conventional resistance training program. Participants will be randomly assigned to one of two groups: (i) a control group performing a conventional home-based resistance training program, (ii) an experimental group following the same program, with the addition of specific long-length eccentric contractions integrated into lower limb exercises.

This trial is designed to address two primary research questions:

(i) Does the integration of long-length eccentric contractions enhance the functional benefits of a conventional resistance training program?

(ii) Are any observed functional improvements associated with specific neuromechanical adaptations?

The corresponding hypotheses are:

1. A home-based resistance training incorporating specific long-length eccentric contractions is more effective to improve functional abilities of healthy old adults.
2. These greater functional improvements result from specific neuromechanical adaptations.

Thirty healthy older adults will be recruited to participate in the study. Initial screening will be conducted via telephone to assess eligibility based on inclusion and exclusion criteria. If concerns arise during this call-specifically, if the participant answers "yes" to any item from the ICOPE Step 1 questionnaire-they will undergo further evaluation by a geriatrist to confirm eligibility. Written informed consent will be obtained from all participants prior to enrollment. Participants will then be semi-randomly allocated to one of two groups: a conventional resistance training group or an experimental group incorporating long-length eccentric contractions, with group assignment stratified to ensure an equal number of men and women in each group. Each participant will complete three laboratory-based experimental sessions and 24 semi-supervised, home-based training sessions over a period of 8 to 11 weeks.

Three experimental sessions will be conducted in the laboratory at the following time points: (i) four weeks prior to training (Pre1), (ii) one week before training (Pre2), and (iii) within one week following the final training session (Post). The two pre-training sessions (Pre1 and Pre2) will establish baseline values for all outcome measures and allow assessment of natural variability in the absence of an intervention. These baseline variations will be compared between groups to ensure initial comparability and to serve as internal controls.

To evaluate training effectiveness, post-training outcomes will be compared between groups using ANCOVA, with Pre2 values as covariates. This approach will directly address the primary research question: Does the addition of long-length eccentric contractions to a conventional training program enhance functional improvements in older adults?

The sessions will consist of 5 evaluations/tests:

5 Time Sit to Stand test, which is the main outcome Timed Up and Go test Measurements of isometric and dynamic muscle strength of the knee extensors and plantar flexors Measurement of cross-sectional areas of vastus lateralis and rectus femoris, as well as gastrocnemius medialis and soleus muscles Measurement of tendon stiffness

At the end of the second experimental session (Pre2), immediately prior to the start of the training intervention, each participant will complete a familiarization session with a researcher, during which they will be guided through the exercises specific to their assigned group (conventional or long-length eccentric program). This session ensures that participants can perform the exercises safely and correctly at home.

Participants will be provided with a training logbook to document their sessions throughout the intervention. They will also receive all necessary equipment, including a weighted vest and a lifting strap, and for those in the long-length eccentric group, an adjustable step platform. To further support autonomy and adherence, participants will be given instructional materials, including video demonstrations and a printed exercise manual.

The intervention will consist of 24 training sessions over a period of 8 to 11 weeks. Of these, 20 sessions will be performed independently at home, while 4 sessions will take place in the laboratory in small groups, supervised by a qualified adapted physical activity instructor and/or physiotherapist.

To maintain engagement and provide support, a researcher will conduct weekly follow-up phone calls to monitor progress, address any questions, and ensure adherence to the training protocol.

Eight different exercises will be included in the training program of both groups, 4 centered around the upper limbs and 4 for the lower limbs:

biceps curls military press triceps extension rowing heel drop: performed on the floor for the conventional group, and performed on the edge of a step for the other group chair squat drop: performed on the floor for the conventional group, and performed with the feet propped up on a step for the other group band dorsiflexion stair descent

Each training session will start with a warm-up and end with a cool-down consisting of stretching and active mobilization (neck, shoulders, elbows, wrists, hips, knee and ankles). The four lower limbs exercises and two upper limbs exercises will be performed each training session, the lower limbs exercises alternating each session between the four given exercises. The intensity of the exercises will be progressively increased by either modifying the execution of the movement (e.g., adjusting step height to alter muscle length) or adding weights, up to a maximum of 20% of the participant' bodyweight. This progression in intensity will be carefully controlled and managed using the CR10 Rating of Perceived Exertion scale. Training volume (calculated as the number of repetitions × number of sets per exercise, in arbitrary units) will gradually increase throughout the training protocol.

During the protocol, participants will be asked not to alter their usual daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 60 years and older
* Individuals eligible for social security coverage
* Individuals without health issues (e.g., musculoskeletal injuries, chronic conditions)
* Individuals who have given their informed consent

Exclusion Criteria:

* Accustomed to resistance exercise (i.e., no participation in a resistance training program within the 6 months prior to enrollment, or not engaging in lower-limb resistance training more than once per week as part of their current routine).
* Pathologies affecting muscle strength in the lower limbs (e.g., neurological or neuromuscular conditions, history of ankle or knee trauma)
* Individuals residing in a healthcare or social institution
* Individuals receiving psychiatric care
* Individuals deprived of their liberty
* Adults under legal protection (guardianship, curatorship, or legal safeguard)
* Participation in another ongoing biomedical research study
* Individuals in an emergency situation
* Individuals not covered by social security
* BMI over 30
* Minimal Mental State Examination (MMSE) score of 25 or lower
* Significant visual impairment

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
5 times Sit to Stand | At baseline (i.e., prior to the start of training) and at study completion (i.e., within one week following the final training session
  The subjects will complete five times STS repetitions on a standardized armless chair. After the cue "ready, set, go!", the subjects will start performing STS repetitions as rapidly as possible from the sitting position with their buttocks touching the chair to the full standing position, with their arms crossed over the chest. Verbal encouragement will be given during the test. The STS test will finish when the subjects sit on the chair after the fifth STS repetition, and the time needed to complete the task will be recorded with a stopwatch to the nearest 0.01 s.

SECONDARY OUTCOMES:
Isometric and dynamic muscle strength | At baseline (i.e., prior to the start of training) and at study completion (i.e., within one week following the final training session
  Participants will be seated on an isokinetic ergometer with hips at 70° and knees at 80° flexion (0° = full extension). They will perform a warm-up of 5 knee extensions at increasing effort (50-90%). Then, they will perform two isometric and two eccentric maximal voluntary contractions (MVCs) from 0° to 120° of knee flexion at 60°/s.
  Next, in a supine position with knee fully extended and ankle neutral (0°), the same warm-up will be performed for plantar flexion, followed by two isometric MVCs. Ankle passive range of motion will be assessed by moving the foot until stretch-related pain occurs; the maximal dorsiflexion angle will define the range limit. The starting position will be set to ensure a constant 60° range. Then, participants will perform two eccentric MVCs across the full ankle range at 30°/s.
  Strong verbal encouragement will be given throughout. All measurements will be taken on the right side only.
Timed Up and Go Test | At baseline (i.e., prior to the start of training) and at study completion (i.e., within one week following the final training session
  Participants will start seated in a chair with their back against the backrest. At the signal, they will stand up, walk 3 meters as quickly and safely as possible, cross the marked line, turn around, walk back to the chair, and sit down. The timer will start when they begin to rise from the chair and stop when they are seated again.
Cross sectional areas of vastus lateralis (VL), rectus femoris (RF), soleus (SOL) and gastrocnemius medialis (GM) muscles. | At baseline (i.e., prior to the start of training) and at study completion (i.e., within one week following the final training session
  All ultrasound assessments will be conducted by an experienced operator using the Aixplorer Ultimate system (SuperSonic Imagine, France).
  For VL and RF muscles, participants will lie supine, knees extended, feet at bed edge, ankles neutral. Femur length will be defined as the distance between the greater trochanter and lateral femoral condyle. Skin will be marked at 30%, 50%, and 70% of this length. In panoramic mode, transverse images will be recorded at each mark, with the probe moving slowly from RF medial to VL lateral border.
  For MG and SOL muscles, participants will lie prone in the same foot/knee position. Muscle-tendon junctions and femoral condyles will be located to define muscle length. Skin will be marked at 30%, 50%, and 70% of MG and SOL lengths. Panoramic transverse images will be taken at each mark, with the probe moving from medial to lateral border in a slow, controlled, low-pressure sweep.
Stiffness of VL and Achilles tendons | At baseline (i.e., prior to the start of training) and at study completion (i.e., within one week following the final training session
  MG and VL myotendinous junctions displacement will be determined during the isometric contractions using B-mode ultrasound. An echo-absorptive marker will be placed on the skin under the probe to act as a fixed reference from which relative measures of displacement will be calculated with a Matlab script.
  Achilles and VL tendon force will be calculated from the knee and ankle joint moments measured with the isokinetic ergometer and the respective moment arm length taken from MRI studies.
  The tendon force-elongation relationships will be fitted with second-order polynomial functions forced through zero. Tendon stiffness (in N/mm) will be calculated from the slope of a linear fit between 60 and 100 % MVC.
Training metrics | Participants will complete the questions after each training session, resulting in 24 recordings.
  Each participant will receive a training booklet in which they will be asked to report information regarding the adherence, feasibility, and acceptability of the training program, with higher score representing better outcomes. Each parameter will be evaluated through a "yes/no" question or a visual analog scale.

CONTACTS AND LOCATIONS:
Locations (1):
- MIP Laboratory, Nantes University, Nantes, France

IPD SHARING:
Plan to Share IPD: Yes
The Individual Participant Data (IPD) will be made available to other researchers upon request, under specific conditions. A data-sharing plan will be developed in accordance with the relevant ethical guidelines, ensuring participant confidentiality and data protection. We will collaborate with other researchers interested in neuromechanical adaptations and aging-related functional capacities, sharing anonymized data via a secure platform. Access to the IPD will be granted only to those who meet the criteria for research use and will be subject to institutional review board approval. Our intention is to promote transparency and foster further exploration in this field while respecting participant privacy and the integrity of the data.
  We are committed to making the following data available: Study Protocol, Statistical Analysis Plan, Informed Consent Form, and Analytic Code. This will ensure transparency, reproducibility, and facilitate further research in the field
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of study completion.

REFERENCES:
- [Background] Tsai LL, McNamara RJ, Moddel C, Alison JA, McKenzie DK, McKeough ZJ. Home-based telerehabilitation via real-time videoconferencing improves endurance exercise capacity in patients with COPD: The randomized controlled TeleR Study. Respirology. 2017 May;22(4):699-707. doi: 10.1111/resp.12966. Epub 2016 Dec 19. PMID 27992099
- [Background] Thiebaud RS, Funk MD, Abe T. Home-based resistance training for older adults: a systematic review. Geriatr Gerontol Int. 2014 Oct;14(4):750-7. doi: 10.1111/ggi.12326. Epub 2014 Aug 11. PMID 25109883
- [Background] Souron R, Nosaka K, Jubeau M. Changes in central and peripheral neuromuscular fatigue indices after concentric versus eccentric contractions of the knee extensors. Eur J Appl Physiol. 2018 Apr;118(4):805-816. doi: 10.1007/s00421-018-3816-0. Epub 2018 Feb 6. PMID 29411127
- [Background] Schoenfeld BJ, Ogborn DI, Vigotsky AD, Franchi MV, Krieger JW. Hypertrophic Effects of Concentric vs. Eccentric Muscle Actions: A Systematic Review and Meta-analysis. J Strength Cond Res. 2017 Sep;31(9):2599-2608. doi: 10.1519/JSC.0000000000001983. PMID 28486337
- [Background] Marusic J, Vatovec R, Markovic G, Sarabon N. Effects of eccentric training at long-muscle length on architectural and functional characteristics of the hamstrings. Scand J Med Sci Sports. 2020 Nov;30(11):2130-2142. doi: 10.1111/sms.13770. Epub 2020 Jul 30. PMID 32706442
- [Background] Maeo S, Huang M, Wu Y, Sakurai H, Kusagawa Y, Sugiyama T, Kanehisa H, Isaka T. Greater Hamstrings Muscle Hypertrophy but Similar Damage Protection after Training at Long versus Short Muscle Lengths. Med Sci Sports Exerc. 2021 Apr 1;53(4):825-837. doi: 10.1249/MSS.0000000000002523. PMID 33009197
- [Background] LaStayo PC, Pierotti DJ, Pifer J, Hoppeler H, Lindstedt SL. Eccentric ergometry: increases in locomotor muscle size and strength at low training intensities. Am J Physiol Regul Integr Comp Physiol. 2000 May;278(5):R1282-8. doi: 10.1152/ajpregu.2000.278.5.R1282. PMID 10801298
- [Background] Katsura Y, Takeda N, Hara T, Takahashi S, Nosaka K. Comparison between eccentric and concentric resistance exercise training without equipment for changes in muscle strength and functional fitness of older adults. Eur J Appl Physiol. 2019 Jul;119(7):1581-1590. doi: 10.1007/s00421-019-04147-0. Epub 2019 May 4. PMID 31055678
- [Background] Guex K, Degache F, Morisod C, Sailly M, Millet GP. Hamstring Architectural and Functional Adaptations Following Long vs. Short Muscle Length Eccentric Training. Front Physiol. 2016 Aug 3;7:340. doi: 10.3389/fphys.2016.00340. eCollection 2016. PMID 27536252
- [Background] Fitze DP, Franchi MV, Muller Brusco C, Engeler N, Frey WO, Sporri J. Hamstrings and quadriceps muscle size and strength in female and male elite competitive alpine skiers. Front Physiol. 2025 Jan 9;15:1444300. doi: 10.3389/fphys.2024.1444300. eCollection 2024. PMID 39850451
- [Background] Doguet V, Nosaka K, Guevel A, Thickbroom G, Ishimura K, Jubeau M. Muscle length effect on corticospinal excitability during maximal concentric, isometric and eccentric contractions of the knee extensors. Exp Physiol. 2017 Nov 1;102(11):1513-1523. doi: 10.1113/EP086480. Epub 2017 Sep 30. PMID 28796385
- [Background] Doguet V, Jubeau M, Dorel S, Couturier A, Lacourpaille L, Guevel A, Guilhem G. Time-Course of Neuromuscular Changes during and after Maximal Eccentric Contractions. Front Physiol. 2016 Apr 18;7:137. doi: 10.3389/fphys.2016.00137. eCollection 2016. PMID 27148075
- [Background] Clarke EC, Martin JH, d'Entremont AG, Pandy MG, Wilson DR, Herbert RD. A non-invasive, 3D, dynamic MRI method for measuring muscle moment arms in vivo: demonstration in the human ankle joint and Achilles tendon. Med Eng Phys. 2015 Jan;37(1):93-9. doi: 10.1016/j.medengphy.2014.11.003. Epub 2014 Nov 26. PMID 25466777
- [Background] Bizet B, Nordez A, Tallio T, Lacourpaille L, Cattagni T, Colard J, Betus Y, Dorel S, Sarcher A, Seynnes O, Andrade RJ. Eight weeks of eccentric training at long-muscle length increases fascicle length independently of adaptations in passive mechanical properties. J Appl Physiol (1985). 2025 Apr 1;138(4):939-949. doi: 10.1152/japplphysiol.00859.2024. Epub 2025 Mar 6. PMID 40048648
- [Background] Blazevich AJ, Coleman DR, Horne S, Cannavan D. Anatomical predictors of maximum isometric and concentric knee extensor moment. Eur J Appl Physiol. 2009 Apr;105(6):869-78. doi: 10.1007/s00421-008-0972-7. Epub 2009 Jan 20. PMID 19153760
- [Background] Chaabene H, Prieske O, Herz M, Moran J, Hohne J, Kliegl R, Ramirez-Campillo R, Behm DG, Hortobagyi T, Granacher U. Home-based exercise programmes improve physical fitness of healthy older adults: A PRISMA-compliant systematic review and meta-analysis with relevance for COVID-19. Ageing Res Rev. 2021 May;67:101265. doi: 10.1016/j.arr.2021.101265. Epub 2021 Feb 8. PMID 33571702
- See also: Website — https://anr-emule.com